CLINICAL TRIAL: NCT06638983
Title: Effectives of Non-extraction Orthodontic Treatment of Angle Class I Malocclusion: A Non-randomized Pre-post Interventional Study
Brief Title: Effectives of Non-extraction Orthodontic Treatment of Angle Class I Malocclusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Can Tho University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ChauHongDiemCtump
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2020-05

CONDITIONS: Angle Class I
Keywords: Non-extraction; orthodontics treatment; Angle class I malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class I

STUDY DESIGN:
Intervention Model Description: Cephalometric radiographs, and extraoral and intraoral photographs, and cast impressions were collected before and after intervention. The weighted PAR Index (Peer Assessment Rating) employed to determine outcome of orthodontic treatment. Also the following soft tissue and bone indexes were assessed before and after intervention, SNA, SNB, ANB, SN_GoGn, SN_Occplane, U1_NAmm, U1_NA, L1_NBmm, L1_NB, U1_L1, U1_Mp, Ls_E, Li_E, and Nasolabial_angle. Intervention was MBT (MBT System, 3M Unitek, USA) non-extraction fixed orthodontic treatment. One experienced researcher analyzed and interpreted all of the cephalometric images used in the study using the WedCeph (https://webceph.com/). Data were analyzed by linear regression and T-Test statistical test using R software version 4.3.0 (R Foundation for Statistical Computing, Vienna, Austria) by a blinded statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cephalometric radiographs and cast impressions were collected before and after intervention. (Other): Cephalometric radiographs, and extraoral and intraoral photographs, and cast impressions were collected before and after intervention. The weighted PAR Index (Peer Assessment Rating) employed to determine outcome of orthodontic treatment.
  Interventions: Other: Non-extraction Orthodontic Treatment of Angle Class I Malocclusion

INTERVENTIONS:
Other: Non-extraction Orthodontic Treatment of Angle Class I Malocclusion — Cephalometric radiographs, and extraoral and intraoral photographs, and cast impressions were collected before and after intervention. The weighted PAR Index (Peer Assessment Rating) employed to determine outcome of orthodontic treatment. Also the following soft tissue and bone indexes were assessed before and after intervention

SUMMARY:
Introduction: The investigators aimed to evaluate the effectiveness of non-extraction orthodontic treatment for Angle class I malocclusion.

DETAILED DESCRIPTION:
Many people are also concerned about their oral health. When social communication is more important, aesthetic concerns also receive a lot of attention. A beautiful smile can boost self-assurance and empathy. Angle class I malocclusion is prevalent, and dental malocclusion is a significant percentage of the population at all ages . Tooth extraction is a controversial topic in orthodontics, with the general view being against it. Angle and his students argued against it, but Charles Tweed saw recurrence in the 1930s after retreatment without extraction and retreatment with extraction. The use of tooth extraction therapy increased in the 1960s but has become less common since the late 20th century. The science of orthodontics has made significant advancements under the principle of least invasiveness, but the debate remains about whether to consider tooth extraction. The contemporary view believes that the majority of patients may and should be treated without tooth extraction, but in rare circumstances, extraction is necessary to make up for crowding and excessive incisor protrusion that harm the beauty. In truth, each individual must be thoroughly evaluated in light of their bite, cosmetic condition, and stability in the wake of therapy before any course of action is recommended. The investigators aimed to evaluate the effectiveness of non-extraction orthodontic treatment for Angle class I malocclusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients (≥ 15 years) with indicated Angle class I malocclusion and missing space ≤9mm
* Cervical vertebral maturation stages 5, 6, (CS5, CS6): cervical vertebrae 2, 3, and 4 have a concave curved lower border and have at least one rectangle C3, C4 cervical vertebra upright or at least square
* No prior orthodontic treatment
* Fully erupted permanent teeth (except third molars)
* Voluntary research participation

Exclusion Criteria:

Face soft tissue surgical procedures, periodontal disease, and maxillofacial congenital anomalies

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
We aimed to evaluate the effectiveness of non-extraction orthodontic treatment for Angle class I malocclusion. | Cephalometric radiographs, and extraoral and intraoral photographs, cast impressions and PAR Index (Peer Assessment Rating) were collected before and after intervention through study completion, an average of 2 years
  Cephalometric radiographs, and extraoral and intraoral photographs, and cast impressions were collected before and after intervention. The weighted PAR Index (Peer Assessment Rating) employed to determine outcome of orthodontic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Diem Chau Hong, DDS, Principal Investigator — Can Tho University of Medicine and Pharmacy
Locations (1):
- Can Tho University of Medicine and Pharmacy, Can Tho, Vietnam

REFERENCES:
- [Result] Baik KM, Anbar G, Alshaikh A, Banjar A. Effect of Social Media on Patient's Perception of Dental Aesthetics in Saudi Arabia. Int J Dent. 2022 Feb 27;2022:4794497. doi: 10.1155/2022/4794497. eCollection 2022. PMID 35265132